CLINICAL TRIAL: NCT03558451
Title: Effectiveness of a Sexual Health Intervention in Women With Genitourinary Syndrome of Menopause to Improve Their Quality of Life. Multicentre Clinical Trial. Project EXIMe
Brief Title: Multicentre Clinical Trial. Project EXIMe
Acronym: EXIMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Fundación de Innovación e Investigación Biomédica de Atención Primaria-Madrid (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCI 24/16
Record Dates: First submitted 2018-02-05; First posted 2018-06-15 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2019-08

CONDITIONS: Menopause
Keywords: Primary health care
MeSH Terms: interventions — Sexual Health

STUDY DESIGN:
Intervention Model Description: Multicentre randomized clinical trial with groups in parallel, controlled single-blind, with blind evaluation of the response variable, held in the Community of Madrid
Who Masked: Participant, Outcomes Assessor
Masking Description: Only primary care midwives know and apply the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXIMe intervention (Experimental): In addition to the usual assistance, women will receive a complex intervention in sexual health, individualized, in the midwife consultation, where techniques for expression, analysis, information and development of sexual health skills will be used.
  Interventions: Other: Complex intervention in sexual health; Other: Usual care
- Usual care (Active Comparator): Usual care according to available protocols applicable to the women and the health service standardized portfolio
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Complex intervention in sexual health — EXIMe is a complex intervention in sexual health, individualized, in the midwife consultation, where techniques for expression, analysis, information and development of sexual health skills will be used.
  Other Names: Usual care
  Arms: EXIMe intervention
Other: Usual care — According to available protocols applicable to the patient and the health service standardized portfolio
  Other Names: Women will receive the usual assistance

SUMMARY:
Objective: to evaluate the effectiveness of an individualized intervention in sexual health conducted in the midwife consultation to improve the quality of life in women with Genitourinary Syndrome of Menopause. Design: Multicentre randomized clinical trial with groups in parallel, controlled single-blind, with blind evaluation of the response variable, held in the Community of Madrid.

DETAILED DESCRIPTION:
Genitourinary Syndrome of Menopause is a common condition that increases by four the risk of having a sexual dysfunction, and that affects the quality of life of women who suffer it. Those women with an active sexual life have fewer symptoms associated with this syndrome. Objective: to evaluate the effectiveness of an individualized intervention in sexual health conducted in the midwife consultation to improve the quality of life in women with Genitourinary Syndrome of Menopause. Design: Multicentre randomized clinical trial with groups in parallel, controlled single-blind, with blind evaluation of the response variable, held in the Community of Madrid. Population: women aged between 45-65 years with Genitourinary Syndrome of Menopause attending to the midwife consultation. N= 250 (125 women in each group) will be included by midwifes in the Primary Health Care consultations in the Community of Madrid. Control group: women will receive the usual assistance.

Experimental group: in addition to the usual assistance, women will receive a complex intervention in sexual health, individualized, in the midwife consultation, where techniques for expression, analysis, information and development of sexual health skills will be used. Variables: Main-Quality of life in menopause (measured with the Cervantes Short-Form Scale). Secondary- sociodemographic variables, sexual history and variables related to the Genitourinary Syndrome of Menopause. Analysis: by intention-to-treat, comparing the quality of life in menopause scores before/after the intervention in both groups after 0, 1 and 6 months. To explain the factors associated with a higher quality of life, a linear regression model would be fitted.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 45-65 years with Genitourinary Syndrome of Menopause

Exclusion Criteria:

* women who present pathologies that lead to an alteration of sexual desire
* women who receive or have received in the last six months treatment that increase the incidence of vaginal atrophy
* women who receive or have received local hormonal therapy during the last month, systemic hormonal therapy in the last six months, or other systemic treatment for the Genitourinary Syndrome of Menopause
* women who could not read or write, and not understand the spanish language.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Main-Quality of life in menopause | Change from baseline Quality of life at six months
  Main-Quality of life in menopause measured with "Cervantes Short-Form Scale" (20 -100 points)

SECONDARY OUTCOMES:
Sexual function | Change from baseline at six months
  Sexual function: measured with Questionnaire "Health and female sexual dysfunction in primary care"
vaginal pH | Change from baseline at six months
  vaginal pH
Oxford scale | Change from baseline at six months
  Oxford scale: pelvic floor muscle response
Urine sediment | Change from baseline at six months
  Urine sediment

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Martinez-Villarejo, Midwife, Principal Investigator — Gerencia de Atención Primaria, Madrid
Locations (1):
- Gerencia de Atención Primaria, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No